CLINICAL TRIAL: NCT04882956
Title: Outcome of Brolucizumab-dbll and Aflibercept Intravitreal Injection in the Treatment of Age-related Macular Neovascular Degeneration
Brief Title: BEOVU Versus Eylea in the Treatment of Age-related Macular Neovascular Degeneration
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Tarek Roshdy mohamed Mahgoub ELhamaky, Professor (associate), Benha University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Hamaky11
Record Dates: First submitted 2021-05-06; First posted 2021-05-12 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2021-05

CONDITIONS: Macula Lutea Degeneration
Keywords: macular degeneration; BEOVU; Eylea
MeSH Terms: conditions — Macular Degeneration | interventions — Intravitreal Injections; aflibercept

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BEOVU (Active Comparator): Intravitreal injection of BEOVU 3 loading injections ( monthly) then every 3 months
  Interventions: Drug: intravitreal injection
- Eylea (Active Comparator): Intravitreal injection of Eylea 3 loading injections ( monthly) then every 3 months
  Interventions: Drug: intravitreal injection

INTERVENTIONS:
Drug: intravitreal injection — Brolucizumab-Dbll intravitreal injection
  Other Names: BEOVU
  Arms: BEOVU
Drug: intravitreal injection — Aflipercept intravitreal injection
  Other Names: Eylea
  Arms: Eylea

SUMMARY:
Age-Related macular neovascularization degeneration occur is a vision threatening condition. The investigators compare the efficacy of BEOVU and Eylea intravitreal treatment in the management.

DETAILED DESCRIPTION:
Baseline ,and postoperative 1 ,6 and 12 months full ophthalmic examination was done. Procedure included randomized intravitreal injection of Brolucizumab (BEOVU®, Genentech, South Francisco, CA) and of aflibercept (Eylea; Regeneron, Tarrytown,NY)

ELIGIBILITY:
Inclusion Criteria:

* • Age-Related macular neovascularization degeneration

Exclusion Criteria:

* other causes of macular neovascularization degeneration
* other macular diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-08-05 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Best corrected visual acuity (BCVA) | 12 months
  Change in BCVA in LOG MARS(logarithm minimum angle of resolution

CONTACTS AND LOCATIONS:
Overall Officials: Tarek Elhamaky, MD, Principal Investigator — Benha University
Locations (1):
- INMC, Abu Dhabi, United Arab Emirates

IPD SHARING:
Plan to Share IPD: Yes
by direct contact through email
Supporting Information: Study Protocol, SAP
Time Frame: unlimited
Access Criteria: direct request by email